CLINICAL TRIAL: NCT07221227
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, 3-Arm Study to Investigate the Safety and Efficacy of Efimosfermin Alfa in Participants With Biopsy-Confirmed F2- or F3-Stage Metabolic Dysfunction-Associated Steatohepatitis (MASH) (ZENITH-1)
Brief Title: A Pivotal Clinical Study to Investigate Efimosfermin Alfa in Participants With Biopsy-confirmed F2- or F3-stage MASH
Acronym: ZENITH-1
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 301160; 2025-523675-39 (Other: EU CT Number)
Record Dates: First submitted 2025-10-15; First posted 2025-10-27 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Non-alcoholic Fatty Liver Disease
Keywords: Efimosfermin Alfa; Metabolic Dysfunction-Associated Steatohepatitis; Non-alcoholic Fatty Liver Disease; ZENITH-1
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This is a double blind study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Participants receiving dose level 1 of efimosfermin alfa (Experimental)
  Interventions: Drug: Efimosfermin alfa
- Participants receiving dose level 2 of efimosfermin alfa (Experimental)
  Interventions: Drug: Efimosfermin alfa
- Participants receiving Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Efimosfermin alfa — Efimosfermin alfa will be administered
  Arms: Participants receiving dose level 1 of efimosfermin alfa
Drug: Efimosfermin alfa — Efimosfermin alfa will be administered
  Arms: Participants receiving dose level 2 of efimosfermin alfa
Drug: Placebo — Placebo will be administered
  Arms: Participants receiving Placebo

SUMMARY:
The purpose of this study is to assess the safety and efficacy of efimosfermin alfa in the resolution of steatohepatitis and improvement of liver-related clinical outcome compared to placebo in individuals with MASH and biopsy-confirmed F2- or F3-stage fibrosis.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to understand and sign a written informed consent form that must be obtained prior to the initiation of study procedures
2. Age >=18 and <=75 years at enrollment
3. History or presence of 2 or more of the 5 components of metabolic syndrome per American Heart Association definition:
4. Liver biopsy confirmation of MASH consistent with stage F2 or F3 fibrosis and a NAS score >=4 confirmed by a central pathologist

Exclusion Criteria:

1. Contraindication or ineligibility for percutaneous liver biopsy
2. ALT or AST >=5*upper limit of normal (ULN)
3. Total bilirubin (BILI) >=1.3 milligram per deciliter (mg/dL). Individuals with documented Gilbert's syndrome may be enrolled if they experienced an isolated increase in total BILI of >=1.3 mg/dL and direct BILI is <=20% of total BILI; otherwise, the individual will be excluded.
4. Serum albumin <=3.5 grams per deciliter (g/dL)
5. International normalized ratio (INR) >=1.3 not due to therapeutic anticoagulation. Individuals receiving chronic anticoagulant treatment with higher INR values may be enrolled at the discretion of the Investigator and Study Medical Monitor.
6. Alkaline phosphatase (ALP) >=2*ULN
7. Platelet (PLT) count <140,000 per (/) cubic millimeter (mm^3); individuals with a PLT count between 110,000/mm^3 and 140,000/mm^3 may be enrolled after discussion with the Study Medical Monitor.
8. Serum creatinine >=1.5 mg/dL or creatinine clearance <=60 milliliter (mL)/minute (min)/1.73 square meter by Chronic Kidney Disease Epidemiology Collaboration equation
9. Alpha-fetoprotein >=20 nanogram per milliliter (ng/mL)
10. Glycated hemoglobin >=9.0%
11. Model for End-Stage Liver Disease score >=12 unless the score is elevated in the absence of liver dysfunction (e.g., Gilbert's syndrome)
12. Phosphatidyl ethanol (PEth) >=80 ng/mL at Screening
13. Known co-infection with any of the following:

    1. Human immunodeficiency virus;
    2. Hepatitis B virus;
    3. Hepatitis C virus (HCV);
    4. Hepatitis D virus; or
    5. Hepatitis E virus.
14. Chronic liver disease from any other cause including, but not limited to, alcoholic liver disease; evidence of portal hypertension; viral hepatitis or any history or evidence of cirrhosis on screening liver biopsy; or decompensated liver disease such as clinical ascites, bleeding gastroesophageal varices, hepatorenal syndrome, or hepatic encephalopathy prior to Screening or Day 1.
15. Current or history of excessive alcohol intake for >=3 months within the 12-month period prior to Screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2025-10-23 (Actual); Primary Completion 2028-03-29 (Estimated); Study Completion 2031-12-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants experiencing improvement in fibrosis by >=1 stage and no worsening of steatohepatitis at Week 52 | At Week 52
  Proportion of participants experiencing improvement in fibrosis of greater than or equal to (>=) 1 stage by MASH clinical research network (CRN) fibrosis scores and no worsening of steatohepatitis (defined as no increase in nonalcoholic fatty liver disease activity score [NAS] for ballooning, inflammation, or steatosis) at 52 weeks will be assessed. MASH CRN fibrosis score ranges from 0 to 4, higher score indicates greater severity. NAS score ranges from 0 to 8, higher score indicates worse disease activity.
Proportion of participants experiencing resolution of steatohepatitis reading and no worsening of MASH CRN fibrosis score at Week 52 | At Week 52
  Resolution of steatohepatitis is defined as absence of fatty liver disease or isolated or simple steatosis without steatohepatitis and a NAS of 0 or 1 for inflammation, 0 for ballooning, and any value for steatosis. NAS score ranges from 0 to 8, higher score indicates worse disease activity. MASH CRN fibrosis score ranges from 0 to 4, higher score indicates greater severity.
Time from randomization to an adjudicated composite liver-related clinical outcome | From Randomization (Day 1) to 48 months
  Liver-related outcome will be comprised of all-cause mortality; transplantation; occurrence of significant hepatic events..

SECONDARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs) and TEAEs by severity | At Week 52 and at Month 48
Number of participants with TEAEs leading to discontinuation and TEAEs leading to discontinuation by severity | At Week 52 and at Month 48
Number of participants with Grade 3 and Grade 4 laboratory abnormalities | At Week 52 and at Month 48
Proportion of participants experiencing resolution of steatohepatitis on overall histopathological reading and improvement in liver fibrosis of >=1 stage at Week 52 | At Week 52
  Resolution of steatohepatitis is defined as absence of fatty liver disease or isolated or simple steatosis without steatohepatitis on overall histopathological reading on liver biopsies. Proportion of participants experiencing improvement in fibrosis of >=1 stage by MASH CRN fibrosis scores and resolution of steatohepatitis on overall histopathological reading at 52 weeks will be assessed. MASH CRN fibrosis score ranges from 0 to 4, higher score indicates greater severity
Proportion of participants experiencing improvement in fibrosis by >=1 stage and no worsening of Steatohepatitis at Month 48 | At Month 48
  Proportion of participants experiencing improvement in fibrosis of >=1 stage by MASH CRN fibrosis scores and no worsening of steatohepatitis (defined as no increase in NAS for ballooning, inflammation, or steatosis) at Month 48 will be assessed. MASH CRN fibrosis score ranges from 0 to 4, higher score indicates greater severity. NAS score ranges from 0 to 8, higher score indicates worse disease activity.
Proportion of participants experiencing improvement in fibrosis by >=2 stage and no worsening of Steatohepatitis at Week 52 and Month 48 | At Week 52 and Month 48
  Proportion of participants experiencing improvement in fibrosis of >=2 stage by MASH CRN fibrosis scores and no worsening of steatohepatitis (defined as no increase in NAS for ballooning, inflammation, or steatosis) at at Week 52 and Month 48 will be assessed. MASH CRN fibrosis score ranges from 0 to 4, higher score indicates greater severity. NAS score ranges from 0 to 8, higher score indicates worse disease activity
Proportion of participants experiencing resolution of steatohepatitis reading and no worsening of MASH CRN score at Month 48 | At Month 48
  Resolution of steatohepatitis is defined as absence of fatty liver disease or isolated or simple steatosis without steatohepatitis and a NAS of 0 or 1 for inflammation, 0 for ballooning, and any value for steatosis. NAS score ranges from 0 to 8, higher score indicates worse disease activity. MASH CRN fibrosis score ranges from 0 to 4, higher score indicates greater severity.
Absolute change from Baseline in vibration-controlled transient elastography-liver stiffness measurement (VCTE-LSM) | Baseline (Day 1), Week 52 and Month 48
Percent Change from Baseline in VCTE-LSM | Baseline (Day 1), Week 52 and Month 48
Absolute change from Baseline in controlled attenuation parameter (CAP) scores | Baseline (Day 1), Week 52 and Month 48
  The CAP score is measured by FibroScan, will be used to quantify and detect liver fat. CAP less than (<) 238 decibel-milliwatts (dB/m) indicated no hepatic steatosis, 238 less than or equal to (<=) CAP <=259 dB/m denoted mild steatosis, 260 <=CAP <=291 dB/m indicated moderate steatosis, and CAP greater than (>) 291 dB/m denoted severe steatosis.
Percent Change from Baseline in CAP scores | Baseline (Day 1), Week 52 and Month 48
  The CAP score is measured by FibroScan, will be used to quantify and detect liver fat. CAP <238 dB/m indicated no hepatic steatosis, 238 <=CAP <=259 dB/m denoted mild steatosis, 260 <=CAP <=291 dB/m indicated moderate steatosis, and CAP >291 dB/m denoted severe steatosis.
Proportion of participants achieving Change from Baseline in VCTE-LSM >=30 percent (%) at Week 52 and Month 48 | Baseline (Day 1), Week 52 and Month 48
  VCTE-LSM is a non-invasive test that uses vibration-controlled transient elastography to measure the stiffness of the liver in kilopascal (kPa).
Absolute change from Baseline in magnetic resonance elastography (MRE) scores | Baseline (Day 1), Week 52 and Month 48
  MRE is a non-invasive imaging technique that combine magnetic resonance imaging (MRI) scanning with low-frequency mechanical vibrations to measure the stiffness of liver. MRE scores <2.5 is normal, 2.5 - 3.0 Normal or inflammation, 3.0 - 3.5 Stage 1-2 fibrosis, 3.5 - 4.0 Stage 2-3 fibrosis, 4.0 - 5.0 Stage 3-4 fibrosis and > 5.0 Stage 4 fibrosis.
Percent Change from Baseline in MRE Score | Baseline (Day 1), Week 52 and Month 48
  MRE is a non-invasive imaging technique that combine MRI scanning with low-frequency mechanical vibrations to measure the stiffness of liver. MRE scores <2.5 is normal, 2.5 - 3.0 Normal or inflammation, 3.0 - 3.5 Stage 1-2 fibrosis, 3.5 - 4.0 Stage 2-3 fibrosis, 4.0 - 5.0 Stage 3-4 fibrosis and > 5.0 Stage 4 fibrosis.
Absolute change from Baseline in Enhanced Liver Fibrosis (ELF) Score | Baseline (Day 1), Week 52 and Month 48
  The ELF score will be calculated using a published algorithm combining the values of a set of extracellular matrix markers. The ELF score is used as a prognostic marker for disease progression: ELF score <9.8: Low risk of progression, ELF score 9.8 to <11.3: Moderate risk of progression and ELF score >=11.3: High risk of progression.
Percent Change from Baseline in ELF Score | Baseline (Day 1), Week 52 and Month 48
  The ELF score will be calculated using a published algorithm combining the values of a set of extracellular matrix markers. The ELF score is used as a prognostic marker for disease progression: ELF score <9.8: Low risk of progression, ELF score 9.8 to <11.3: Moderate risk of progression and ELF score >=11.3: High risk of progression.
Proportion of participants experiencing improvement in ELF score of >=0.5 | At Week 52 and Month 48
  The ELF score will be calculated using a published algorithm combining the values of a set of extracellular matrix markers. The ELF score is used as a prognostic marker for disease progression: ELF score <9.8: Low risk of progression, ELF score 9.8 to <11.3: Moderate risk of progression and ELF score >=11.3: High risk of progression.
Absolute change from Baseline in hepatic fat fraction (HFF) by MRI-derived proton density fat fraction (PDFF) | Baseline (Day 1), Week 52 and Month 48
  HFF is the percentage of fat in the liver measured by MRI proton density fat fraction technique, which ranges from 0-75%. Greater than 5% is considered extra fat in the liver.
Percent Change from Baseline in HFF by MRI-PDFF | Baseline (Day 1), Week 52 and Month 48
  HFF is the percentage of fat in the liver measured by MRI proton density fat fraction technique, which ranges from 0-75%. Greater than 5% is considered extra fat in the liver.
Absolute change from Baseline in alanine aminotransferase (ALT) and aspartate aminotransferase (AST) (International units per liter) | Baseline (Day 1), Week 52 and Month 48
Percent Change from Baseline in ALT and AST (International units per liter) | Baseline (Day 1), Week 52 and Month 48
Absolute change from Baseline in ALT and AST ratio (ALT/AST) | Baseline (Day 1), Week 52 and Month 48
  ALT/AST ratio is calculated as ALT/AST ratio equal to ALT divided by AST.
Percent Change from Baseline in ALT and AST ratio (ALT/AST) | Baseline (Day 1), Week 52 and Month 48
  ALT/AST ratio is calculated as ALT/AST ratio equal to ALT divided by AST.
Proportion of participants experiencing ALT and HFF normalization at Week 52 and Month 48 | At Week 52 and Month 48
Proportion of participants experiencing HFF <=5% at Week 52 and Month 48 | At Week 52 and Month 48
  HFF is the percentage of fat in the liver measured by MRI proton density fat fraction technique, which ranges from 0-75%. Less than or equal to 5% is considered normal (no significant fatty infiltration (steatosis) in the liver.
Change from Baseline in glycated hemoglobin (HbA1c) (Percentage of HbA1c) in participants with Type 2 Diabetes Mellitus (T2DM) | Baseline (Day 1), Week 52 and Month 48
Change from Baseline in body weight (kilograms) | Baseline (Day 1), Week 52 and Month 48
Change from Baseline in fasting total cholesterol, low-density lipoprotein (LDL)-cholesterol, high-density lipoprotein (HDL)- cholesterol, and triglycerides (Millimoles per liter) | Baseline (Day 1), Week 52 and Month 48
Proportion of participants with antidrug and antiFGF21 antibody (ADA) | At Week 52 and Month 48
Change from Baseline in Chronic Liver Disease Questionnaire-Nonalcoholic Steatohepatitis (CLDQ-NASH) in domain and total score | Baseline (Day 1), Week 52 and Month 48
  CLDQ-NASH is a NASH-specific health-related quality of life (HRQoL) Patient-Reported Outcomes (PRO) designed to assess 6 health domains over 36 items: abdominal symptoms (3 items), activity/energy (5 items), emotional health (9 items), fatigue (6 items), systemic symptoms (6 items) and worry (7 items). The domain scores range from 1 to 7, higher scores indicating better HRQoL. A score of 1 meaning the symptom being assessed is "present always" while a score of 7 means the symptom is "never present". The total score can range from 36 to 252, a higher score corresponds to a better quality of life while a lower score corresponds to a worse quality of life.
Change from Baseline in Short Form-36 (SF-36) component and domain scores at Week 52 and Month 48 | Baseline (Day 1), Week 52 and Month 48
  SF-36 is a generic HRQoL PRO designed to assess 8 health domains over 36 items: physical functioning (10 items), bodily pain (2 items), role limitations due to physical problems (4 items), role limitations due to emotional problems (3 items), general health (5 items), mental health (5 items), social functioning (2 items), and vitality (4 items). Each domain is scored from 0 (poorer health) to 100 (better health). SF-36 is scored into 8 domains and 2 component scores: physical component summary (PCS) and mental component summary (MCS). The domain and component scores range from 0 to 100, with higher scores indicating better HRQoL.
Serum drug Concentration of efimosfermin alfa | Up to Month 48
Maximum serum drug concentration (Cmax) of efimosfermin alfa | Up to Month 48
Area under the serum concentration-time curve (AUC) of efimosfermin alfa | Up to Month 48
Average serum drug concentration (Cavg) of efimosfermin alfa | Up to Month 48
Serum concentration of study drug at the end of the dosing interval (Ctrough) of efimosfermin alfa | Up to Month 48
Exposure-response relationship for efimosfermin alfa | Baseline (Day 1), Week 52 and Month 48
  To evaluate the correlation between pharmacokinetics (PK) derived from plasma concentrations, and biomarker responses, safety, and efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Study Sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or asset(s) with development terminated across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf